CLINICAL TRIAL: NCT07159607
Title: Positron Emission Tomography-based Response Assessment in Isocitrate Dehydrogenase (IDH)-Mutant Gliomas - a Bicentric, Prospective, Observational Study
Brief Title: Amino Acid PET-based Response Assessment in IDH-mutant Gliomas (APPEAR)
Acronym: APPEAR
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Servier Affaires Médicales (Industry); Servier Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Nathalie Albert, Prof. Dr. med., LMU Klinikum
Other Study IDs: 24-1114
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: IDH-mutant Glioma (Oligodendroglioma, Astrocytoma)
Keywords: APPEAR; PET-basierte Beurteilung des Therapieansprechens in Isocitrat-Dehydrogenase (IDH)-mutierten Gliomen - eine prospektive Beobachtungsstudie; Isocitrate dehydrogenase mutant gliomas; Positron emission tomography; FET PET; PET RANO; Amino acid PET; glioma
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The radiological follow-up of diffuse gliomas is challenged by the difficult distinction of true progression from treatment-related changes. To this end, the Response Assessment in Neuro-Oncology (RANO) Working Group has issued specific recommendation for the standardized evaluation of magnetic resonance imaging (MRI). In addition, positron emission tomography (PET) using radiolabeled amino acids allows for the delineation of metabolically active tumor regions in brain tumors, and guidelines for PET-based response assessment have been recently proposed (PET RANO 1.0). However, well-annotated data on longitudinal PET alterations before and during treatment and follow-up are missing in isocitrate dehydrogenase (IDH)-mutant gliomas, particularly as tumor entities defined by IDH mutations have been established only recently and data on PET imaging mainly rely on previous brain tumor classification frameworks.

Aims: This bicentric, prospective, observational study aims to collect data on imaging-based disease monitoring in patients with IDH-mutant gliomas. Specifically, this study aims to investigate longitudinal changes of amino acid PET tracer uptake during treatment in IDH-mutant gliomas and to evaluate the correlation between amino acid PET uptake at baseline and response to postoperative standard of care treatment.

Patient cohort/methods: Adult (age ≥ 18 years) patients diagnosed and/or treated at the Medical University of Vienna (Vienna, Austria) or the LMU Hospital Munich (Munich, Germany) with histologically verified diffuse IDH-mutant glioma (oligodendroglioma, astrocytoma of all grades) and PET imaging for routine follow-up before, during and after treatment will be included. Clinical and imaging data will be collected in a standardized manner and correlated with treatment response. Primary endpoint is progression-free survival (PFS) according to RANO 2.0 criteria, secondary endpoints include PFS according to PET-RANO 1.0 criteria, time to next intervention (TTNI) and overall survival (OS).

Originality/relevance: This study will generate data that will inform future response assessment frameworks and the design of future clinical trials in IDH-mutant glioma.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Histologically verified diffuse IDH-mutant glioma (astrocytoma, oligodendroglioma) of any grade as defined in the WHO classification of tumors of the central nervous system
* Postoperative treatment according to current standard of care at the time of study inclusion
* Performance of amino acid PET as part of clinical routine

Exclusion Criteria:

* Inclusion in another clinical trial/investigational study involving an experimental therapy or study medication
* Inclusion criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age ≥ 18 years) patients diagnosed and/or treated at the Medical University of Vienna (Vienna, Austria) or the LMU Hospital Munich (Munich, Germany) with histologically verified diffuse IDH-mutant glioma (oligodendroglioma, CNS WHO grades 2 and 3; astrocytoma, CNS WHO grades 2, 3 and 4) and PET imaging for routinely performed response assessment before, during and after first-line treatment will be included after obtaining informed consent. In total, we expect the inclusion of 100 patients over an accrual period of 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2030-07-16 (Estimated); Study Completion 2030-07-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From enrollment at least 24 months, maximal until end of study (max. 24 months after enrolment of last patient).
  PET image information at baseline and follow-up as well as responses according to PET RANO 1.0 criteria will be correlated with progression-free survival (PFS) according to RANO 2.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie L Albert, Prof. Dr. med., Principal Investigator — LMU Klinikum München
Locations (2):
- Medical University of Vienna, Vienna, Austria
- LMU Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be considered upon reasonable request, depending on ethics approval